CLINICAL TRIAL: NCT06959303
Title: The Effect of Discharge Training With Teach-Back Method on Anxiety, Fear of Death and Knowledge Level in Patients Undergoing Coronary Angiography: A Randomised Controlled Study
Brief Title: Effect of Teach-Back Method in Angiography
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Asst. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TarsusU-NBARISEREN-003
Record Dates: First submitted 2025-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Angiography
Keywords: Angiography; teach-back; anxiety; fear of death; knowledge level; education
MeSH Terms: conditions — Anxiety Disorders; Necrophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach back education group (Experimental): In the first stage, all participants will be explained about the research and their consent will be obtained. 'Personal Information Form' will be filled out for the patients whose informed consents are obtained and who agree to participate in the study. Then, 'Information Questionnaire', 'State Anxiety Scale' and 'Death Anxiety Scale' will be administered to all patients as a pretest. In the second stage, discharge training will be given to patients who underwent coronary angiography with the Teach-Back method. In the third stage, 'Information Questionnaire', 'State Anxiety Scale' and 'Death Anxiety Scale' will be applied as posttest after the training. In addition, at the end of the study, 'Satisfaction Evaluation of Teach-Back Method' will be made to the intervention group.
  Interventions: Behavioral: Teach Back Education
- Control Group (No Intervention): In the first stage, all participants will be explained about the research and their consent will be obtained. 'Personal Information Form' will be filled out for the patients whose informed consents are obtained and who agree to participate in the study. Then, 'Information Questionnaire', 'State Anxiety Scale' and 'Death Anxiety Scale' will be administered to all patients as a pretest. No intervention will be made in the second stage. The routine process in the hospital will continue. In the third stage, 'Information Questionnaire', 'State Anxiety Scale' and 'Death Anxiety Scale' will be applied as posttest.

INTERVENTIONS:
Behavioral: Teach Back Education — Discharge training will be given to patients who underwent coronary angiography with the Teach-Back method.
  Arms: Teach back education group

SUMMARY:
This study aims to evaluate the effect of discharge training with Teach-Back Method on anxiety, fear of death and knowledge level in patients undergoing coronary angiography.

H1: The training given with the Teach-Back Method decreases the anxiety level of coronary angiography patient.

H2: The training given with the Teach-Back Method decreases the fear of death level of coronary angiography patient.

H3: The training given with the Teach-Back Method increases the knowledge level of coronary angiography patient.

DETAILED DESCRIPTION:
Teach-back technique is an effective educational method that enables a person to rephrase what he/she has learnt in his/her own words to show that he/she understands. There is no study evaluating the effect of discharge training with Teach-Back Method on anxiety, fear of death and knowledge level in patients undergoing coronary angiography. In addition, in this study, anxiety, fear of death and knowledge levels of the patients before and after the training will be discussed and will guide future studies. Discharge education to be given with the Teach-Back method will increase the level of knowledge of the patients and enable them to return to their normal lives. At the end of the study, the participants will be asked about their satisfaction level with the Teach-Back method. According to the results of the study, it is expected that the use of the Teach-Back method will increase in the education given to patients.

ELIGIBILITY:
Inclusion Criteria:

* To have the ability to communicate verbally,
* Volunteering to participate in the research,
* To be 18 years of age or older.

Exclusion Criteria:

* Lack of verbal communication skills,
* Not volunteering to participate in the research,
* Being under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 10 minutes
  This form was prepared by the researchers in line with the literature and includes questions questioning the demographic characteristics such as age, gender, socioeconomic level, etc. This form will be used before the training.
Information Questionnaire | 20 minutes
  This form will consist of questions that will measure the level of knowledge of patients about discharge education after coronary angiography. A literature review will be conducted and 20 multiple-choice questions will be prepared by the researchers. Expert opinion will be obtained from a total of 5 faculty members working in the department of nursing principles in the preparation of this form. Then, the form will be finalised after the necessary arrangements are made. In the form consisting of multiple-choice questions with one correct answer, each question has a value of 5 points. Caregivers can get at least 0 and at most 100 points from the knowledge test. Increasing the score means that the knowledge is sufficient. Questions with incorrect answers are considered as topics to be prioritised in training. This form will be used before and after the training.
State Anxiety Inventory | 10 minutes
  This scale was developed by Spielberger and colleagues (1970). The scale was adapted into Turkish by Öner and Le Compte (1998). The scale consists of 20 questions and it is a scale that determines how the individual feels at a certain moment and condition. In the state anxiety scale, the response options collected in four classes are: (1) Not at all, (2) A little, (3) A lot and (4) Completely. The constant value for the State Anxiety Scale is 50. The scores obtained in the state anxiety scale theoretically vary between 20 and 80 points. In the evaluation of the scale, it is accepted that those who score below 36 have no anxiety, those who score between 37 and 42 have mild anxiety and those who score 42 and above have high anxiety. This form will be used before and after the training.
Death Anxiety Scale | 10 minutes
  This scale was developed by Templer (1970). The scale was adapted into Turkish by Şenol (1989). The validity and reliability of this scale was reviewed by Akça and Köse (2008) in different groups in Turkish norms.The scale consists of 15 items expressing feelings such as anxiety, fear, and terror related to death. The scale is in the form of true and false binary Likert type. Correct answers are given 1 point, while incorrect answers are not scored. In the test with a score range of 0-15, a higher score means that death anxiety is higher. It can be said that those with a scale score of 7 and above also have high death anxiety. This form will be used before and after the training.
Evaluation of Satisfaction with Teach-Back Method | 5 minutes
  The patients participating in the study will be asked to give a score between 1-10 in order to determine the level of satisfaction with the training provided by the teach-back method. It is defined as 1-not at all 10- very much and they will be asked to give full points. This form will be used after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen D, Huang W, Wei S, Zhu Y, Shi B. The impact of Teach-back method on preoperative anxiety and surgical cooperation in elderly patients undergoing outpatient ophthalmology surgery: A randomized clinical trial. Medicine (Baltimore). 2023 Feb 22;102(8):e32931. doi: 10.1097/MD.0000000000032931. PMID 36827029
- [Background] Oh S, Choi H, Oh EG, Lee JY. Effectiveness of discharge education using teach-back method on readmission among heart failure patients: A systematic review and meta-analysis. Patient Educ Couns. 2023 Feb;107:107559. doi: 10.1016/j.pec.2022.11.001. Epub 2022 Nov 4. PMID 36411152
- [Background] Oh EG, Lee JY, Lee HJ, Oh S. Effects of discharge education using teach-back methods in patients with heart failure: A randomized controlled trial. Int J Nurs Stud. 2023 Apr;140:104453. doi: 10.1016/j.ijnurstu.2023.104453. Epub 2023 Feb 4. PMID 36827745
- [Background] Oh EG, Lee HJ, Yang YL, Kim YM. Effectiveness of Discharge Education With the Teach-Back Method on 30-Day Readmission: A Systematic Review. J Patient Saf. 2021 Jun 1;17(4):305-310. doi: 10.1097/PTS.0000000000000596. PMID 30882616
- [Background] Cutilli CC. Excellence in Patient Education: Evidence-Based Education that "Sticks" and Improves Patient Outcomes. Nurs Clin North Am. 2020 Jun;55(2):267-282. doi: 10.1016/j.cnur.2020.02.007. PMID 32389259
- [Background] Huang J, Lin X, Xiong D, Huang K, Luo X, Lin Q, Li M, Zhang P. Impact of the teach-back method on caregiver outcomes using the "Timing it Right" framework for hemodialysis patients. Front Public Health. 2023 Jun 23;11:1123006. doi: 10.3389/fpubh.2023.1123006. eCollection 2023. PMID 37427278
- [Background] Eloi H. Implementing teach-back during patient discharge education. Nurs Forum. 2021 Jul;56(3):766-771. doi: 10.1111/nuf.12585. Epub 2021 Apr 30. PMID 33931873
- [Background] Choi S, Choi J. Effects of the teach-back method among cancer patients: a systematic review of the literature. Support Care Cancer. 2021 Dec;29(12):7259-7268. doi: 10.1007/s00520-021-06445-w. Epub 2021 Jul 24. PMID 34302545
- [Background] Ahmadidarrehsima S, Bidmeshki EA, Rahnama M, Babaei K, Afshari M, Khandani BK. The Effect of Self-Management Education by the Teach-Back Method on Uncertainty of Patients with Breast Cancer: a Quasi-Experimental Study. J Cancer Educ. 2020 Apr;35(2):366-372. doi: 10.1007/s13187-019-1474-5. PMID 30680649